CLINICAL TRIAL: NCT01940016
Title: A Feasibility Study on the Effects of Tailored Communication and Health Coach Support on Physical Activity in Overweight Postmenopausal Women: BePHIT
Brief Title: Communication & Peer Support Effects on Physical Activity in Overweight Postmenopausal Women
Acronym: BePHIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Electra Paskett, Associate Director for Population Sciences, Comprehensive Cancer Center, Ohio State University; Marion N. Rowley Professor of Cancer Research and Director, Division of Cancer Prevention and Control, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-05005; NCI-2012-00204 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-07-13; First posted 2013-09-11 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Healthy; Obesity; Postmenopausal
Keywords: Feasibility study; Interactive voice response system (IVR); health coach; no evidence of disease
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (health coach) (Experimental): Participants participate in a 12-week physical activity intervention (walking program)and receive health mail messages via IVR system and from a health coach. Participants in this arm of the study, interacted with the IVR system and had the option of interacting with the health coach.
  Interventions: Behavioral: communication intervention; Behavioral: exercise intervention
- Arm II (no coach condition) (Active Comparator): Participants participate in a 12-week physical activity intervention (walking program)and receive health mail messages via IVR system. Participants in this arm of the study only interacted with the IVR system.
  Interventions: Behavioral: exercise intervention

INTERVENTIONS:
Behavioral: communication intervention — Participants participate in a 12-week physical activity intervention (walking program)and receive health mail messages via IVR system and had the option of communicating with a health coach.
  Arms: Arm I (health coach)
Behavioral: exercise intervention — Participants participate in a 12-week physical activity intervention administered using an IVR system.

SUMMARY:
This randomized clinical trial studies the feasibility of tailored physical activity intervention that is administered using Interactive Voice Response technology and cell phones. Interactive voice response and health coach support may motivate overweight postmenopausal women to stick to their exercise regimen to reduce the risk of getting breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To design, develop and test the feasibility of implementing a physical activity intervention using tailored communication and Interactive Voice Response (IVR) technology. We will to address four basic questions to accomplish this aim:

1. Among overweight, postmenopausal women, who pass the screening criteria, what is the percentage of women who are willing to participate in a 12-week physical activity intervention that includes two 1-mile walk tests and two visits to the General Clinical Research Center (GCRC)?
2. After beginning the study, what proportion of women use the cell phone and land line at least 5 days a week to get a physical activity intervention message?
3. How many participants are enrolled and participating in the study at the end of the 12-week intervention period?
4. On average, how many steps per day do participants walk? How many of the participants reach the 10,000 steps-per-day target by the end of the 12 week-intervention?

SECONDARY OBJECTIVES:

I. The effectiveness (satisfaction, convenience, ease of operation) of all the materials and processes.

II. Examine whether social support from a health coach results in improvements in our measures of adherence and satisfaction.

III. Examine the correlation between self-reported steps per day with improvements in performance on a 1-mile walk test administered at the beginning and the end of the 12-week intervention.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I. COACH-CONDITION: Participants participate in a 12-week physical activity program (walking program)and receive health mail messages via IVR system and from a health coach. Participants in this arm of the study, interacted with the IVR system and had the option of interacting with the health coach.

ARM II: NO-COACH CONDITION: Participants participate in a 12-week physical activity program (walking program) administered using an IVR system.

ELIGIBILITY:
Inclusion Criteria:

* Present a letter/documentation from a primary physician stating that they can participate in a physical activity program that will require walking up to 10,000 steps per day
* Have a body mass index (BMI) between 25 and 40 kg/m^2 (inclusive)
* Be postmenopausal, defined as no period for 12 months if over age 55, or no period for 12 months; also, women who have had their ovaries removed will be considered as postmenopausal
* Willing to participate in a wellness program that lasts 12 weeks and involves walking for at least 30 minutes a day on most days
* Has access to a cell phone during the 12-week intervention
* Functional knowledge of English (ability to both read and write)

Exclusion Criteria:

* Taking hormone replacement therapy within 3 months of enrollment
* Taking Tamoxifen or Raloxifene within 3 months of enrollment
* Enrolled in a weight management program, such as Weight Watchers
* Engaged in regular, planned walking of at least 30 minutes a day
* Previous history of breast cancer
* Premenopausal
* Age > 75 years, to minimize co-morbidities
* Cannot walk one mile

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2009-11-01 (Actual); Study Completion 2009-11-01 (Actual)

PRIMARY OUTCOMES:
Change in time taken to complete a one mile walk. | 12 weeks

SECONDARY OUTCOMES:
Changes in anthropometrics, psychometrics and the benefits of a health coach. | 12 weeks
Weekly effectiveness (satisfaction, convenience, ease of operation) of all the materials and processes as assessed by questionnaires. | 12 weeks
If the self-reported steps per day, derived from daily activity logs, relates to the change in performance on the 1-mile walk test between baseline and end of study. | 12 Week
  The steps walked per day and the change in performance on the 1-male walk test are both outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Electra Paskett, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu